CLINICAL TRIAL: NCT03799510
Title: Safety and Immunogenicity Evaluation of the Vaccine Candidate Sm14 Against Schistosomiasis in Senegalese School Children Healthy or Infected With S. Mansoni and/or S. Haematobium. A Comparative, Randomized, Controlled, Open-label Trial
Brief Title: Anti-Schistosomiasis Vaccine: Sm14 Phase 2b-Sn in School Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Orygen Biotecnologia SA (Unknown); Biomedical Research Center EPLS (Other); Access to Advanced Health Institute (AAHI) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sm14 Phase 2b - Sn
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Schistosomiasis
Keywords: Schistosomiasis; Recombinant vaccine; rSm14; GLA-SE; Fatty acid-binding protein (FABP); Phase II Clinical Trial; Senegal
MeSH Terms: conditions — Schistosomiasis | interventions — SM14 protein, Schistosoma mansoni; glucopyranosyl lipid-A

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Healthy school children with no infectious history of Schistosomiasis receiving three (3) intramuscular injections of 50 μg Sm14 with 2.5 μg GLA-SE solution at D0, W4, W8 (D=day; W=week). Three-month follow-up (W12, W20).
  Interventions: Biological: Sm14; Drug: GLA-SE solution
- Group 2 (Experimental): School children with an infectious history of S. haematobium and-or S. mansoni and pretreated with 1 dose of Praziquantel (2-4 weeks prior to the first vaccine injection) receiving three (3) intramuscular injections of 50 μg Sm14 with 2.5 μg GLA-SE solution at D0, W4, W8 (D=day; W=week). Three-month follow-up (W12, W20).
  Interventions: Biological: Sm14; Drug: GLA-SE solution
- Group 3 (No Intervention): School children with an infectious history of S. haematobium and S. mansoni and pretreated with 1 dose of Praziquantel (2-4 weeks prior to the first vaccine injection) not receiving vaccine. Control group.

INTERVENTIONS:
Biological: Sm14 — Three 0.5 mL intra-muscular injections of the vaccine solution (50μg Sm14) will be administered on D0, W4, W8 (D = day, W = week).
  Other Names: rSm14
  Arms: Group 1; Group 2
Drug: GLA-SE solution — The lot concentration 10μg/mL for injection of 2.5μg GLA-SE/injection.
  Other Names: • Glucopyranosyl Lipid A in Stable Emulsion; • Glucopyranosyl Lipid Adjuvant-Stable Emulsion; • Toll-like Receptor 4 Agonist GLA-SE
  Arms: Group 1; Group 2

SUMMARY:
The clinical trial phase 2b is designed to assess the safety and the specific immune response of the active ingredient (protein + adjuvant) in healthy and then in infected school children from 8 to 11 years of age with intestinal and/or urinary schistosomiasis, living in the Valley of the Senegal River, a highly endemic area for schistosomiasis.

DETAILED DESCRIPTION:
A phase 2b trial, self-contained, open-label, controlled, randomized study in three parallel arms, two of them formed by groups of healthy or infected school children, both receiving three (3) injections at D0, W4 (Week 4), W8; both groups receiving 50 μg Sm14 vaccine candidate solution, combined with 2.5μg GLA-SE. The third group is composed by non-vaccinated infected school children.

Sm14: recombinant protein produced in yeast following Good Manufacturing Practices (GMP) conditions, presented in vials containing 0.55 ml solution Sm14, 0.4 ml solution is diluted with 0.4 ml of GLA (Synthetic Glucopyranosyl lipid A) for intramuscular administration.

Medical examinations are performed at D0 (before injection, 1 hr and 4 hr after), and a safety evaluation at 24 hrs and 48 hrs, after each injection.

Blood analysis: Liver function tests - renal function tests - blood counts, at W-1 before inclusion, and at W9 and W21 during the follow-up.

Blood samples for immune response analysis at D0, W12 and W21.

ELIGIBILITY:
Inclusion Criteria:

* School children, of public schools in villages of Saint Louis region (Senegal), female or male, 8 to 11 years old (inclusive) at the time of inclusion.
* Residence in the area during the period of the study.
* Free of obvious/severe health problems except schistosomiasis, as established by clinical examination.
* Written informed consent to participate obtained from subject's parents or legal guardian.
* Free of obvious/severe health problems except schistosomiasis, established by blood analysis, i.e. hematological exams, liver and renal function tests.
* Treated with 40mg/kg Praziquantel (PZQ) before inclusion (W-2 to W-4 before the first injection) in case of infection with S. mansoni and S. haematobium
* Children of Group 1: not infected, no schistosomiasis history and living in area/village free of Sm and Sh transmission.
* Children Groups 2 & 3: infected with mansoni or/and haematobium schistosomiasis.

Exclusion Criteria:

* School child who does not respond to one of the inclusion criteria
* Child under 20kg of body weight
* Vaccination within 90 days preceding the first dose of Sm14 vaccine candidate, or planned use during the study period.
* Current or previous chronic administration (defined as more than 14 days) of immunosuppressive drugs or other immuno-modifying drugs.
* Known hypersensitivity to any component in the Sm14 vaccine or history of allergic disease.
* Knowledge of non-infectious chronic disease
* Known acute disease.
* Other conditions which in opinion of the PI may potentially represent a danger for the patient to be enrolled.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | within 2 days of the administration of the first dose (Day 0)
  Local signs and symptoms included Pain, Swelling and Inflammation at the injection site, heaviness or pain upon passive or active movement of the injected limb, Complete physical examination including an examination of general appearance, body weight and forehead temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates.
  General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day 30-Day 32: within 2 days of the administration of the second dose (Week 4)
  Local signs and symptoms included Pain, Swelling and Inflammation at the injection site, Heaviness or pain upon passive or active movement of the injected limb, Complete physical examination including an examination of general appearance, body weight and forehead temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates.
  General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Days 60-67 : within 7 days of the administration of the third dose (Week 8)
  Local signs and symptoms included Pain, Swelling and Inflammation at the injection site. Heaviness or pain upon passive or active movement of the injected limb, Complete physical examination including an examination of general appearance, body weight and forehead temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates.
  General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances. Laboratory tests (blood count, liver and kidney biological functions).
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day 90: three months after the first injection (Week 12)
  Injection local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection. Complete physical examination including an examination of general appearance, body weight and forehead temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day 120: four months after the first injection (Week 16)
  Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection.
  Complete physical examination including an examination of general appearance, body weight and forehead temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day 150: five months after the first injection (Week 21)
  Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection.
  Complete physical examination including an examination of general appearance, body weight and forehead temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances.

SECONDARY OUTCOMES:
Qualitative and quantitative assessment of the Immunogenicity | The Day of first Sm14 vaccine administration (Day 0)
  Immunogenicity was evaluated by Isotype analysis of the antibodies produced specifically against the rSm14 and vaccine-induced (ELISA) and Specific rSm14 cellular response (on PBMC), production of intracellular cytokines (PBMCs stimulation and cytokine dosing). Cellular immune responses measured by PBMC luminex assay for T-cell cytokines (Milliplex ® MAP kit).
  Correlation between the development and magnitude of humoral responses measured by antibody IgG production to the Sm14 Schisto protein using enzyme-linked immunosorbent assay (ELISA).
Qualitative and quantitative assessment of the Immunogenicity | At the 30th day after the third Sm14 vaccine administration (Week 12)
  Immunogenicity was evaluated by Isotype analysis of the antibodies produced specifically against the rSm14 and vaccine-induced (ELISA) and Specific rSm14 cellular response (on PBMC), production of intracellular cytokines (PBMCs stimulation and cytokine dosing). Cellular immune responses measured by PBMC luminex assay for T-cell cytokines (Milliplex ® MAP kit).
  Correlation between the development and magnitude of humoral responses measured by antibody IgG production to the Sm14 Schisto protein using enzyme-linked immunosorbent assay (ELISA).
Qualitative and quantitative assessment of the Immunogenicity | At the 90th day after the third Sm14 vaccine administration (Week 21)
  Immunogenicity was evaluated by Isotype analysis of the antibodies produced specifically against the rSm14 andvaccine-induced (ELISA) and Specific rSm14 cellular response (on PBMC), production of intracellular cytokines (PBMCs stimulation and cytokine dosing). Cellular immune responses measured by PBMC luminex assay for T-cell cytokines (Milliplex ® MAP kit).
  Correlation between the development and magnitude of humoral responses measured by antibody IgG production to the Sm14 Schisto protein using enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Tendler, MD, PhD, Study Chair — Oswaldo Cruz Foundation; Modou DIOP, MD, Principal Investigator — Biomedical Research Center ESPOIR POUR LA SANTE (BRC-EPLS); Gilles RIVEAU, PharmD, PhD, Study Director — Biomedical Research Center ESPOIR POUR LA SANTE (BRC-EPLS).; Anne-Marie SCHACHT, CRA, Study Director — Biomedical Research Center ESPOIR POUR LA SANTE (BRC-EPLS).
Locations (1):
- Biomedical Research Center EPLS, Saint-Louis, Senegal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moser D, Tendler M, Griffiths G, Klinkert MQ. A 14-kDa Schistosoma mansoni polypeptide is homologous to a gene family of fatty acid binding proteins. J Biol Chem. 1991 May 5;266(13):8447-54. PMID 2022660
- [Result] Ramos CR, Spisni A, Oyama S Jr, Sforca ML, Ramos HR, Vilar MM, Alves AC, Figueredo RC, Tendler M, Zanchin NI, Pertinhez TA, Ho PL. Stability improvement of the fatty acid binding protein Sm14 from S. mansoni by Cys replacement: structural and functional characterization of a vaccine candidate. Biochim Biophys Acta. 2009 Apr;1794(4):655-62. doi: 10.1016/j.bbapap.2008.12.010. Epub 2008 Dec 25. PMID 19150418
- [Result] Coler RN, Bertholet S, Moutaftsi M, Guderian JA, Windish HP, Baldwin SL, Laughlin EM, Duthie MS, Fox CB, Carter D, Friede M, Vedvick TS, Reed SG. Development and characterization of synthetic glucopyranosyl lipid adjuvant system as a vaccine adjuvant. PLoS One. 2011 Jan 26;6(1):e16333. doi: 10.1371/journal.pone.0016333. PMID 21298114
- [Result] Santini-Oliveira M, Coler RN, Parra J, Veloso V, Jayashankar L, Pinto PM, Ciol MA, Bergquist R, Reed SG, Tendler M. Schistosomiasis vaccine candidate Sm14/GLA-SE: Phase 1 safety and immunogenicity clinical trial in healthy, male adults. Vaccine. 2016 Jan 20;34(4):586-594. doi: 10.1016/j.vaccine.2015.10.027. Epub 2015 Nov 10. PMID 26571311
- [Result] Lambert SL, Yang CF, Liu Z, Sweetwood R, Zhao J, Cheng L, Jin H, Woo J. Molecular and cellular response profiles induced by the TLR4 agonist-based adjuvant Glucopyranosyl Lipid A. PLoS One. 2012;7(12):e51618. doi: 10.1371/journal.pone.0051618. Epub 2012 Dec 28. PMID 23284726
- [Result] Tendler M, Almeida MS, Vilar MM, Pinto PM, Limaverde-Sousa G. Current Status of the Sm14/GLA-SE Schistosomiasis Vaccine: Overcoming Barriers and Paradigms towards the First Anti-Parasitic Human(itarian) Vaccine. Trop Med Infect Dis. 2018 Nov 21;3(4):121. doi: 10.3390/tropicalmed3040121. PMID 30469320